CLINICAL TRIAL: NCT00625248
Title: A Prospective Evaluation of Bleeding Risk of Anticoagulant and Antiplatelet Therapy for Interventional Techniques
Brief Title: Prospective Evaluation of Bleeding Risk of Anticoagulant and Anti-platelet Therapy
Status: Completed | Type: Observational
Sponsor: Pain Management Center of Paducah (Other)
Responsible Party: Principal Investigator, Laxmaiah Manchikanti, MD, Medical Director, Pain Management Center of Paducah
Other Study IDs: protocol 18
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — Anticoagulants; Platelet Aggregation Inhibitors

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- no anthithrombotic: procedures where there were no antithrombotics
  Interventions: Drug: Antithrombotics
- Antithrombotic - continued: patients who are on antithrombotics
  Interventions: Drug: Antithrombotics
- Discontinued Antithrombotic: Patients who were on antithrombotics but have been discontinued
  Interventions: Drug: Antithrombotics

INTERVENTIONS:
Drug: Antithrombotics — With or without or discontinuted use of Antithrombotics
  Other Names: anticoagulant or antiplatelet drugs

SUMMARY:
This study will evaluate bleeding risk and differences in outcomes in patients receiving and not receiving anticoagulant or antiplatelet therapy

DETAILED DESCRIPTION:
1. To evaluate bleeding risk in interventional procedures in patients with or without antiplatelet and/or anticoagulant therapy.
2. To evaluate differences in outcomes in patients not receiving any anticoagulant or antiplatelet therapy compared to patients receiving various types of drugs with anticoagulant or antiplatelet therapeutic effects.
3. To evaluate and compare the adverse event profiling all patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing interventional techniques. Subjects who were able to give voluntary, written informed consent.

Exclusion Criteria:

* All those things, patients on heparin, dextran, and low molecular heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ambulatory surgery center patients
Sampling Method: Probability Sample
Enrollment: 12000 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To evaluate for differences between the patients undergoing interventional techniques with or without anticoagulant or antiplatelet therapy. | 24 months

SECONDARY OUTCOMES:
To assess adverse events in all patients. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Laxmaiah Manchikanti, MD, Principal Investigator — Ambulatory Surgery Center, Paducah
Locations (1):
- Pain Management Center of Paducah, Paducah, Kentucky, United States

REFERENCES:
- [Result] Manchikanti L, Malla Y, Wargo BW, Cash KA, McManus CD, Damron KS, Jackson SD, Pampati V, Fellows B. A prospective evaluation of bleeding risk of interventional techniques in chronic pain. Pain Physician. 2011 Jul-Aug;14(4):317-29. PMID 21785475
- [Derived] Manchikanti L, Malla Y, Wargo BW, Fellows B. Infection control practices (safe injection and medication vial utilization) for interventional techniques: are they based on relative risk management or evidence? Pain Physician. 2011 Sep-Oct;14(5):425-34. PMID 21927046